CLINICAL TRIAL: NCT06897267
Title: The Development and Feasibility of the Peer-based Recovery Program
Brief Title: The Feasibility of the Peer-based Recovery Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: A-ER-112-029
Record Dates: First submitted 2025-03-11; First posted 2025-03-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mental Disorder; Recovery, Psychological
Keywords: peer; recovery program
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Grow to Recovery program-Short Version (Experimental): Intervention group members will receive the Grow to Recovery program -Short version, co-led by one trained peer and one trained professional.
  Interventions: Behavioral: The Grow to Recovery program-Short Version

INTERVENTIONS:
Behavioral: The Grow to Recovery program-Short Version — The program is based on "Pathways to Recovery:A Strengths Recovery Self-help Workbook." After completing the leader training program, one peer and one professional will conduct a 10-week Grow to Recovery program-Short Version for people with mental illness. This program covers recovery concepts, strengths, and goal setting, which will be helpful for people in recovery.

SUMMARY:
Recovery-oriented services are currently the mainstream in the field of mental health around the world. Peer services are an alternative service option promoted by recovery advocates. Western countries have invested abundant resources in promoting peer services and providing training for peer support workers. However, peer services in Taiwan have just started. More resources need to be added to make mental health services catch up with the world trend so that people with mental illness in Taiwan can have more choices. Hence, this study aims to investigate the feasibility of the Grow to Recovery program-Short Version co-led by a peer.

DETAILED DESCRIPTION:
The study will verify the feasibility of the Grow to Recovery program-Short Version co-led by a peer. Based on the previous interview data and related literature, a peer leader training course will be established. One to three peers will be recruited to receive the training, and colead the Grow to Recovery program-Short Version with one trained professional. The pre- and post-test as well as course questionnaire data collected from program participants will be used to establish the feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Professionals:

  1. working in the community psychiatric rehabilitation organizations
  2. being willing to co-lead the recovery program with a peer
* Peers:

  1. having a diagnosis of mental illness over 1 year
  2. living in the community
  3. being age 18 yr or older
  4. having good communication skills
  5. being willing to co-lead the recovery program with a professional
* People with mental illness

  1. having a diagnosis of mental illness over 1 year
  2. living in the community
  3. being age 18 yr or older
  4. filling out the scales independently
  5. being able to participate in a recovery group and follow the group rules

Exclusion Criteria:

* People with mental illness 1. attending another recovery-related group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Stages of Recovery Scale, SRS | Baseline and the 10th week.
  The Stages of Recovery Scale (SRS) consists of 45 items, with six subscales: the sense of hope, disability management/taking responsibility, regaining autonomy, social functioning/role performance, overall well-being, and willingness to help. A higher score means better recovery status.
General Self-Efficacy Scale, GSES | Baseline and the 10th week.
  The General Self-Efficacy Scale (GSES) contains 10 items. A higher score means better self-efficacy.
Medical Outcomes Study Social Support Survey, MOS-SS | Baseline and the 10th week.
  The Medical Outcomes Study Social Support Survey (MOS-SS) is a multidimensional, self-administered instrument that addresses all five functions of an interpersonal relationship to assess the various functional dimensions of social support, including emotional , informational, tangible, affectionate, and positive interaction. A higher score means better social support.
The Hope Scale, THS | Baseline and the 10th week.
  A 12-item Hope Scale (THS) measures the level of sense of hope. A higher score means a higher sense of hope.
Taiwanese Depression Questionnaire, TDQ | Baseline and the 10th week.
  The Taiwanese Depression Questionnaire (TDQ) has 18 items and measures depressed conditions. A higher score means a more depressed mood.
Social Functioning Scale, SFS | Baseline and the 10th week.
  The Social Functioning Scale (SFS) has 36 items. A higher score means better social functioning.
Perceived Psychiatric Stigma Scale, PPSS | Baseline and the 10th week.
  The Perceived Psychiatric Stigma Scale (PPSS) measures self-stigma and has 25 items. A higher score means more severe stigma.

OTHER OUTCOMES:
Course questionnaire | at the end of the intervention (the 10th week)
  The course questionnaire aims to collect course feedback from participants. The questionnaire includes a course-satisfactory survey and open questions. A higher score means higher satisfaction.
Qualitative data | at the end of the intervention (the 10th week)
  The discussion about course feedback in the 10th class will be recorded and transcribed.
Qualitative interview | After completing two cohorts of the Grow to Recovery program-Short Version.
  The researcher will conduct an interview with peer and professional leaders after completing the Grow to Recovery program-Short Version.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ching Chang, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan